CLINICAL TRIAL: NCT01581788
Title: Open Label, Balanced, Randomized, Single-dose, Crossover Oral Bioequivalence Study of Divalproex Sodium ER Tablets 500 mg of Dr. Reddy's and Depakote ER 500 mg Tablets of Abbott Laboratories, in Healthy Subjects Under Fed Conditions.
Brief Title: Bioequivalence Study of Divalproex Sodium ER Tablets, 500 mg Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 10-vin-123
Record Dates: First submitted 2012-04-04; First posted 2012-04-20 (Estimated); Last update posted 2012-04-20 (Estimated); Status verified 2012-04

CONDITIONS: Healthy
Keywords: Bioequivalence; Divalproex Sodium; Crossover
MeSH Terms: interventions — Valproic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Divalproex Sodium ER Tablets, 500 mg (Experimental): Divalproex Sodium ER Tablets, 500 mg of Dr. Reddy's Laboratories Limited
  Interventions: Drug: Divalproex Sodium
- Depakote ER Tablets, 500 mg (Active Comparator): Depakote ER Tablets, 500 mg of Abbott Laboratories
  Interventions: Drug: Divalproex Sodium

INTERVENTIONS:
Drug: Divalproex Sodium — Divalproex Sodium ER Tablets, 500 mg
  Other Names: Depakote

SUMMARY:
The purpose of this study is to assess the bioequivalence between Divalproex Sodium ER Tablets 500 mg of Dr. Reddy's and Depakote ER 500 mg Tablets of Abbott Laboratories in healthy, adult, human subjects, under fed conditions and to monitor adverse events and ensure the safety of subjects.

DETAILED DESCRIPTION:
Open label, balanced, randomized, two-treatment, two-sequence, two-period, single-dose, crossover oral bioequivalence study of Divalproex Sodium Extended Release Tablets 500 mg of Dr. Reddy's Laboratories Limited, and Depakote ER 500 mg mg Tablets of Abbott Laboratories in healthy, adult, human subjects, under fed conditions.

ELIGIBILITY:
Inclusion Criteria:

The subjects were selected for study participation, if they met the following criteria:

1. Subjects aged between 18 and 45 years (both inclusive).
2. Subjects' weight within normal range according to normal values for Body Mass Index (18.5 to 24.9 kg/m2) with minimum of 50 kg weight.
3. Subjects with normal health as determined by personal medical history, clinical examination and laboratory examinations within the clinically acceptable reference range.
4. Subjects having normal 12-lead electrocardiogram (ECG).
5. Subjects having normal chest X-Ray (P/A view) whose X-Ray was taken not more than 6 months prior to the dosing of Period 01.
6. Subjects having negative urine screen for drugs of abuse (including amphetamines, barbiturates, benzodiazepines, marijuana, cocaine, and morphine).
7. Subjects having negative alcohol breath test.
8. Subjects willing to adhere to the protocol requirements and to provide written informed consent.

Exclusion Criteria:

The subjects were excluded from the study, if they met any of the following criteria:

1. Hypersensitivity to Divalproex or related class of drugs.
2. History or presence of significant cardiovascular, pulmonary, hepatic, renal, gastrointestinal, endocrine, immunological, dermatological, neurological or psychiatric disease or disorder.
3. Any treatment which could bring about induction or inhibition of hepatic microsomal enzyme system within 1 month of the study starting.
4. History or presence of significant alcoholism or drug abuse.
5. History or presence of significant smoking (more than 10 cigarettes or beedi's/day).
6. History or presence of asthma, urticaria or other significant allergic reactions.
7. History or presence of significant gastric and/or duodenal ulceration.
8. History or presence of significant thyroid disease, adrenal dysfunction, organic intracranial lesion such as pituitary tumor.
9. History or presence of cancer.
10. Difficulty with donating blood.
11. Difficulty in swallowing solids like tablets or capsules.
12. Use of any prescribed or OTC medication during last two weeks prior to dosing in period 01.
13. Major illness during 3 months before screening.
14. Participation in a drug research study within past 3 months.
15. Donation of blood in the past 3 months before screening.
16. Consumption of grapefruit juice, xanthine-containing products, tobacco containing products or alcohol for within 48 hours prior to dosing.
17. Positive screening test for any one or more: HIV, Hepatitis B and Hepatitis C.
18. History or presence of significant easy bruising or bleeding.
19. History or presence of significant recent trauma.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2011-01; Primary Completion 2011-02 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Area under curve (AUC) | Pre-dose 1 hour, 1.50, 3, 4.50, 6, 7.50, 9, 10.50, 12, 13.50, 15, 16.50, 18, 19.50, 21, 22.50, 24, 25.50, 27, 32, 36, 48, 60, 72, 96 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Gunjan Shah, MBBS, Principal Investigator — Veeda Clinical Research, India
Locations (1):
- Veeda Clinical Research, India, Ahmedabad, Gujarat, India